CLINICAL TRIAL: NCT06959381
Title: Investigation of Acute Effects of Myofascial Release Techniques on Jumping Performance, Balance, and Proprioception in Football Players
Brief Title: Myofascial Release Techniques in Football Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Musa Güneş, Principal Investigator, PhD, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Karabuk-2282
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Fasciae (Anatomy)--Inflammation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fascial release with instrument assisted soft tissue mobilization (Experimental): The fascial release group will be treated with the Graston device to the superficial and deep fascia of the hamstrings and the gastro-soleus muscle complex.
  Interventions: Other: Fascial release with instrument assisted soft tissue mobilization
- Fascial release with foam roller (Experimental): The fascial release group will be treated with the self-foam roller treatment to the fascia of the hamstrings and the gastro-soleus muscle complex.
  Interventions: Other: Fascial release with foam roller
- Control (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: Fascial release with instrument assisted soft tissue mobilization — The fascial release group will be treated with the Graston device to the superficial and deep fascia of the hamstrings and the gastro-soleus muscle complex in both extremities for a total of 16 minutes.
  Arms: Fascial release with instrument assisted soft tissue mobilization
Other: Fascial release with foam roller — Fascial release with a foam roller will be applied to the fascia of the hamstring and gastro-soleus muscle complex with a self-foam roller for a total of 16 minutes.
  Arms: Fascial release with foam roller

SUMMARY:
Fascial tissue ensures optimal function and mobility by providing gliding and force transfer during movement. However, fascial order can be disrupted in cases such as overuse and trauma. Therefore, treatment of fascial tissue is important. Therefore, this study aimed to investigate the effects of different myofascial release techniques on jumping performance, flexibility, balance, and proprioception in amateur football players.

DETAILED DESCRIPTION:
Fascial tissue ensures optimal function by providing gliding and force transfer during movement. It is also associated with an increase in functional capacity by providing flexibility. However, excessive exercise, incorrect movements, and excessive load on the tissue cause dysfunctions in the fascial tissue, leading to myofascial limitations. Elimination of these limitations is important for the maintenance of optimal function. Fascia also provides sensory transmission as a proprioceptive organ. Myofascial limitations also cause problems in sensory organization, leading to injuries and injuries. For this reason, a decrease in flexibility, balance, and sports functions can be observed. Various methods are used to eliminate this myofascial limitation, and there is an increasing demand for myofascial release techniques in many areas daily. The effects of different myofascial release techniques have been examined in the literature in various disease groups and sports injuries, and their effects on joint range of motion, pain, and flexibility have been shown. However, since there are different release techniques, information on which method is more effective or the optimal usage period is unclear. Therefore, this study aimed to investigate the effects of different myofascial release techniques applied with Graston and foam roller on jumping performance, flexibility, balance, and proprioception in amateur football players.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-35
* Being able to communicate in Turkish
* Being willing to participate in the study.
* Being a licensed football player

Exclusion Criteria:

* Those with a body mass index of 30 kg/m² or higher
* Those with a history of lower extremity surgery in the last 6 months
* Those with cardiac, musculoskeletal, vestibular, and neurological problems
* Those with mental, perceptual problems (Mini-mental test score <24)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Jumping perfomance | baseline, immediately after the intervention
  My Jump 2, a mobile app designed for vertical jump performance, high-speed video capture
Proprioception | baseline, immediately after the intervention
  Proprioception will be evaluated with an inclinometer at a 30-45 degree angle.
Balance | baseline, immediately after the intervention
  The Y Balance Test (YBT) will ve used for evaluating dynamic balance across three reach directions: anterior (ANT), posteromedial (PM), and posterolateral (PL)
Flexibilty | baseline, immediately after the intervention
  Flexibility will be assessed with a sit-and-reach test.

CONTACTS AND LOCATIONS:
Overall Officials: Musa Gunes, PhD, Study Director — Karabuk University
Locations (1):
- Karabuk University, Physiotherapy and Rehabilitation Application and Research Center, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] MacDonald GZ, Penney MD, Mullaley ME, Cuconato AL, Drake CD, Behm DG, Button DC. An acute bout of self-myofascial release increases range of motion without a subsequent decrease in muscle activation or force. J Strength Cond Res. 2013 Mar;27(3):812-21. doi: 10.1519/JSC.0b013e31825c2bc1. PMID 22580977
- [Result] Joshi DG, Balthillaya G, Prabhu A. Effect of remote myofascial release on hamstring flexibility in asymptomatic individuals - A randomized clinical trial. J Bodyw Mov Ther. 2018 Jul;22(3):832-837. doi: 10.1016/j.jbmt.2018.01.008. Epub 2018 Feb 17. PMID 30100320
- [Result] Pişirici P, Ekiz MB, İlhan CA. Investigation of the acute effect of myofascial release techniques and dynamic stretch on vertical jump performance in recreationally active individuals. Journal of Physical Education and Sport. 2020;20(3):1569-1579.